CLINICAL TRIAL: NCT02095067
Title: Telemedical Solutions in Medical Emergencies, Advantages and Disadvantages for Patients, Healthcare Professionals, and Healthcare System. Study 2: Videoconferencing Between Ambulances and Physician at the Emergency Medical Dispatch Center,
Brief Title: Videoconferencing Between Ambulances and Physician at the Emergency Medical Dispatch Center, Effects on On-Site Patient Treatment and Patterns of Referral
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Prehospital Medical Emergency Services, Aarhus, Central Denmark Region, Denmark (Unknown); Central Denmark Region (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRAA2
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-03

CONDITIONS: Acute Illness; Acute Injury
Keywords: Telemedicine; Emergency medical dispatch; Prehospital care; Video conference

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Video consultation (Experimental): Patients in this arm receive video consultation from physician at the emergency medical dispatch center
  Interventions: Device: Video consultation
- Telephone consultation (No Intervention): Patients receiving prehospital care by ambulance personnel whom receive telephone consultation/supervision by physician at the emergency medical dispatch center.

INTERVENTIONS:
Device: Video consultation
  Other Names: For video consultation Apple iPad AIR 4G/3G 16GB will be used.; LifeSizeClearSea solution will be used for videoconferencing; 4G/3G mobile network
  Arms: Video consultation

SUMMARY:
The prehospital resources are limited. The emergency medical dispatch center (EMDC) is manned by qualified health care personnel around the clock. The investigators believe that the EMDC is an unexploited resource in the prehospital treatment of patients. By the use of videoconferencing the investigators will activate this resource.

Mobile videoconferencing between ambulances and physician at the EMDC enables patient consultation at a distance. Video consultation between patient and the physician at the EMDC can take place when the patient is at home or in the ambulance.

The primary aim of this study is to examine the effect of video consultation between physicians at the EMDC and patients receiving treatment by ambulance personnel on the number of patients receiving final treatment on-site in the pre hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Less ill/slightly injured patients receiving prehospital care by ambulance personnel

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients receiving final treatment on-site prehospitally | Final treatment is registered for the present consultation, assessed up 36 months, presented up to 36 months

SECONDARY OUTCOMES:
Readmission | Within 3 days of primary contact, assessed up to 36 months, presented up to 36 months
  For all patients receiving consultation from physician at the dispatch center resulting in final treatment on-site, number of patients admitted to hospital within 3 days will be assessed.
Change in site of referral | If destination for patient is changed during consultataion with physician, assessed up to 36 months, presented up to 36 months
  If the department to receive the patient is changed during consultation with physician at the dispatch center.
Number of treatments delivered by ambulance personnel | The number of treatments delivered by ambulance personnel during consultation with physician at the dispatch center, assessed up to 36 months, presented up to 36 months
Change of transportation mode | If mode of transportation is changed during consultation with physician, assessed up to 36 months, presented up to 36 months
  If the mode of transportation is changed during consultation with physician at the dispatch center. Eg. from ambulance to standard patient transportation without monitoring og the possibility of treatment, ether with patient sitting up or lying down.

OTHER OUTCOMES:
Ambulance staff evaluation of usability of equipment | At the time of using the equipment, asessed up to 36 months, presented up to 36 months
  Is investigated by the use of survey
Physicians evaluation of usability of equipment | At the time of using the equipment, assessed up to 36 months, presented up to 36 months
  Is evaluated by the use of survey

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Prehospital Emergency Medical Services, Aarhus, Central Denmark Region, Aarhus N
  - Responce A/S, Horsens